CLINICAL TRIAL: NCT02563249
Title: Influence of Gravity on Dexterity, Hand-eye Coordination and Perception of Orientation and Distances
Acronym: DEXTER0g
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-026
Record Dates: First submitted 2015-07-23; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexterity, Coordination,Perception measurements (Other): Dexterity, Hand-eye Coordination and Perception of Orientation and Distances
  Interventions: Other: Parabolic flight; Other: movements of the upper limb, the gripping force, muscle activity and eye-cephalic subject movement measurements

INTERVENTIONS:
Other: Parabolic flight
Other: movements of the upper limb, the gripping force, muscle activity and eye-cephalic subject movement measurements

SUMMARY:
If investigators know that the anticipatory mechanisms involved in precision grip take into account the gravity, however it is unclear how they adapt to changes in the gravitational level. The objectives of this study are to study and model the movement control and the mechanisms underlying learning and adapting to the condition of weightlessness. Specifically, i) investigators will determine if a change in the level of gravity is taken into account when controlling grip force and ii) investigators will examine the effects of gravity change on hand-eye coordination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male or female
* 18 to 65 years
* Affiliated with a Social Security plan or holder of a European Health Insurance Card (EHIC - European Health Insurance Card - EHIC).
* Having an aeronautical medical certificate of fitness for flight personnel unprofessional functions in civil aviation.
* Agreeing to participate in the study
* Having given informed consent

Exclusion Criteria:

* person not affiliated to a Social Security Inssurance,
* person who participated in a clinical trial within the trial below the exclusion period,
* person with a medical history or any acute or chronic condition that can affect the test results, or by running a risk on during the protocol, especially topics: past or present history of neurological disease, rheumatologic or otologic (hearing or equilibration) OR person with a corrected visual acuity of less than 5 / 10th.
* pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Gravity induced changes in grip strength (newton) exerted between the fingers measured with strain gauges | baseline
Gravity induced changes in oculo-manual coordination measured by the latency (ms) of anticipatory eye movement measurement with videooculography | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France